CLINICAL TRIAL: NCT04490954
Title: A Prospective, Self-paired, Single-center Clinical Trial Evaluating the Accuracy of Brain Biological Electrical Impedance Tomography Screen for Supratentorial Tumors
Brief Title: The Accuracy of Brain Biological Electrical Impedance Tomography Screen for Supratentorial Tumors
Acronym: ABST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IR2019001127
Record Dates: First submitted 2020-07-19; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Brain Tumor; Brain Edema
Keywords: Electrical Impedance Tomography; Supratentorial Brain Tumors
MeSH Terms: conditions — Brain Neoplasms; Brain Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients examined with MRI/CT (Other)
  Interventions: Device: MRI/CT
- Patients examined with biological electrical impedance (Other)
  Interventions: Device: brain biological electrical impedance tomography; Device: MRI/CT

INTERVENTIONS:
Device: brain biological electrical impedance tomography — Patients diagnosed with brain supratentorial tumors through MRI/CT are evaluated with brain biological electrical impedance tomography. And the brain biological electrical impedance tomography is used to monitor the cerebral edema situation of patients with brain edema
  Arms: Patients examined with biological electrical impedance
Device: MRI/CT — Patients diagnosed with brain supratentorial tumors through MRI/CT

SUMMARY:
Compared with MRI or CT, brain biological electrical impedance tomography were performed on patients with supratentorial tumors and healthy people . The AUC (area under the curve) of ROC, which is associated with the increased maximum and the difference between left and right equilibrium of impedance value, is calculated. The specificity of brain biological electrical impedance tomography in screening supratentorial tumors are evaluated.

To compare the changes of parameters detected by brain biological electrical impedance tomography, the enrolled brain tumor patients with cerebral edema were paired with themselves and intravenous infusion of mannitol so that the sensitivity of this device in monitoring cerebral edema can be evaluated.

DETAILED DESCRIPTION:
Compared with MRI or CT, brain biological electrical impedance tomography were performed on patients with supratentorial tumors and healthy people . The AUC (area under the curve) of ROC, which is associated with the increased maximum and the difference between left and right equilibrium of impedance value, is calculated. The specificity of brain biological electrical impedance tomography in screening supratentorial tumors are evaluated.

To compare the changes of parameters detected by brain biological electrical impedance tomography, the enrolled brain tumor patients with cerebral edema were paired with themselves and intravenous infusion of mannitol so that the sensitivity of this device in monitoring cerebral edema can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤70 years old, male or female;
2. Preoperative patients who had been diagnosed with supratentorial tumors by MRI/CT or other conventional methods or healthy people (23 cases each);
3. The longest diameter of the brain tumor is ≥3 cm;
4. Informed Consent Has been signed

Exclusion Criteria:

1. Severe systemic compound injury or hemorrhagic shock;
2. Epilepsy, poisoning symptoms;
3. In critical condition;
4. Patients with brain wounds or acute inflammation;
5. Lactation and pregnant women;
6. Those who have no informed consent ability or cannot sign by themselves;
7. The investigator considers it inappropriate for the patient to participate in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The AUC of ROC curve of the maximum increased value of impedance | 1 year
  The AUC of ROC curve of the maximum increased value of impedance

SECONDARY OUTCOMES:
the difference between the left and right equilibrium | 1 year
  the difference between the left and right equilibrium

CONTACTS AND LOCATIONS:
Overall Officials: 1 year 1 year, M.D., Principal Investigator — Department of neurosurgery
Locations (1):
- Jianmin Zhang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No